CLINICAL TRIAL: NCT06853821
Title: The Effect of Comfort Theory-Based Care and the Use of Virtual Reality Glasses on Pain and Comfort in the Postpartum Period: Randomized Controlled Study
Brief Title: he Effect of Care and the Use of Virtual Reality Glasses on Pain and Comfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-71522473-050.04-363990-135
Record Dates: First submitted 2024-09-03; First posted 2025-03-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Care
Keywords: Postpartum Period; Pain; Comfort Care; Virtual Reality
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were assigned to groups using the "simple randomization" method. Participants were not informed about which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No intervention will be given to the control group.
  Pre-Post Test:
  A personal information form, postpartum comfort scale and visual analog scale will be applied to individuals.
- Experimental Group (Comfort Theory Based Care (Experimental): The experimental group will be intervened by providing comfort theory-based care.
  Pre-Post Test:
  A personal information form, postpartum comfort scale and visual analog scale will be applied to individuals.
  Interventions: Other: Comfort Theory Based Care
- Experimental Group (Virtual Reality Glasses) (Experimental): The experimental group will be intervened with virtual reality glasses.
  Interventions: Other: Virtual Reality Glasses

INTERVENTIONS:
Other: Comfort Theory Based Care — In the research, this group includes care-based intervention
  Arms: Experimental Group (Comfort Theory Based Care
Other: Virtual Reality Glasses — In the research, this group includes interventions with virtual reality glasses.
  Arms: Experimental Group (Virtual Reality Glasses)

SUMMARY:
The research will be conducted to determine the effect of comfort theory-based care and virtual reality glasses on pain and comfort levels in women who have given birth to primiparous babies. The hypotheses of the study are:

H0: Comfort theory-based care and the use of virtual reality glasses have no effect on pain and comfort in the postpartum period.

H1-1: Comfort theory-based care has an effect on pain level in the postpartum period.

H1-2: Comfort theory-based care has an effect on comfort in the postpartum period.

H2-1: The use of virtual reality glasses in the postpartum period has an effect on the level of pain.

H2-2: The use of virtual reality glasses in the postpartum period has an effect on comfort.

DETAILED DESCRIPTION:
Although pregnancy and birth are normal processes, the type of birth affects the comfort level, quality of life, and pain in the natal and postnatal period. In our country, as in many other countries, cesarean delivery rates are quite high.Pain in cesarean births is more severe and lasts longer than in vaginal birth. Along with many methods to reduce pain, the effectiveness of virtual reality applications is also emphasized theoretically or conceptually.In the planned randomized controlled study, the pain level and comfort of individuals will be measured by applying virtual reality glasses to one of the experimental groups and giving Kolcaba's Comfort Theory-based care to the other. Personal Information Form, Postpartum Comfort Scale, Visual Analogue Scale (VAS) and Virtual Reality Glasses Form will be used as measurement tools.This study aims to reduce the pain of the mother in the short term and enable the mother to participate in self-care and baby care in a shorter period of time, and in the long term to minimize maternal and newborn deaths and eliminate deaths under the age of 5.Increasing maternal comfort during the postpartum period is expected to have a direct impact on maintaining maternal health and indirectly on baby care.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Having given birth with epidural anesthesia
* Being between the ages of 18-35
* Having given birth within 37-41 weeks of pregnancy
* Having a primiparous cesarean birth

Exclusion Criteria:

* Having a normal birth
* Having given birth with general anesthesia
* Having a disability that limits vision, hearing or communication
* Having a systemic disease, hypertension, preeclampsia or uterine atony and risk of bleeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Comfort Scale | postpartum first day, postpartum second day, postpartum third day
  It is a 5-point Likert type scale consisting of 34 items developed by Katharine Kolcaba (1994). Cronbach's Alpha number of the scale was determined as 0.78. The minimum score from the scale is 34 and the maximum score is 170. As the score increases, comfort increases.
Visual Analog Scale | postpartum first day, postpartum second day, postpartum third day
  It is used to evaluate pain severity. On the numerical rating scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain) (Huskisson, 1974).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Çevirme, Study Director — acevirme@sakarya.edu.tr
Locations (1):
- Kocaeli State Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolcaba KY. A theory of holistic comfort for nursing. J Adv Nurs. 1994 Jun;19(6):1178-84. doi: 10.1111/j.1365-2648.1994.tb01202.x. PMID 7930099
- [Background] Karakaplan, S. ve Yıldız, H. (2010). Doğum Sonu Konfor Ölçeği geliştirme çalışması. Maltepe Üniversitesi Hemşirelik Bilim ve Sanatı Dergisi, 3(1),55-65.
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420